CLINICAL TRIAL: NCT07103603
Title: Effects of Menopausal Hormone Therapy on Liver Function and Non-Alcoholic Fatty Liver Disease: A Prospective Study
Brief Title: MHT and Liver Function in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ipek B. Ozcivit Erkan, MD (Other)
Responsible Party: Sponsor-Investigator, Ipek B. Ozcivit Erkan, MD, Obstetrician and Gynecologist, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Approval Number:814468
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-07

CONDITIONS: Menopause; Non Alcholic Fatty Liver Disease; Hepatic Steatosis
Keywords: Menopausal hormone therapy; Non-alcoholic fatty liver disease; Liver function; Attenuation imaging; Hepatic steatosis; Postmenopausal women
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease | interventions — Hormone Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: MHT Group (Active Comparator): Postmenopausal women receiving menopausal hormone therapy (oral or transdermal estrogen). Evaluated at baseline and after 6 months for liver function, lipid profile, FIB-4 score, and attenuation imaging.
  Interventions: Drug: Menopausal hormone therapy
- Group 2: Control Group (No Intervention): Postmenopausal women not receiving MHT. Monitored without treatment and evaluated using the same laboratory and imaging parameters.

INTERVENTIONS:
Drug: Menopausal hormone therapy — Menopausal hormone therapy including oral or transdermal estrogen, with or without progestin, administered based on clinical indications.
  Arms: Group 1: MHT Group

SUMMARY:
This prospective study aims to evaluate the effects of menopausal hormone therapy (MHT) on liver function, lipid profiles, and hepatic steatosis in postmenopausal women. A total of 44 participants will be divided into two groups: 22 received MHT and 22 were monitored without treatment. Biochemical parameters, FIB-4 scores, and attenuation imaging (ATI) measurements are assessed at baseline and after six months. The study investigates whether MHT is associated with favorable changes in liver enzymes, hepatic fat accumulation, and noninvasive fibrosis markers.

DETAILED DESCRIPTION:
This prospective, controlled cohort study is designed to evaluate the effects of menopausal hormone therapy (MHT) on liver function and non-alcoholic fatty liver disease (NAFLD) in postmenopausal women. A total of 44 participants are included and divided into two groups: 22 women will receive MHT and 22 will be monitored without treatment due to the absence of menopausal symptoms.

Biochemical parameters including liver enzymes and lipid profiles are measured at baseline and after six months. In addition, hepatic steatosis is quantitatively assessed using attenuation imaging (ATI), a novel ultrasound-based technique, and FIB-4 scores are calculated as noninvasive indicators of liver fibrosis.

The MHT regimens included both oral and transdermal estrogen, selected based on clinical indications. ATI measurements are performed using standardized protocols by radiologists blinded to clinical data.

The primary aim of the study is to investigate whether MHT is associated with favorable changes in hepatic steatosis and liver-related biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 40 years or older
* Postmenopausal status (defined as ≥12 months of amenorrhea)
* No prior use of menopausal hormone therapy in the last 6 months
* Willingness to participate and provide informed consent

Exclusion Criteria:

* History of liver disease, liver malignancy, or liver transplantation
* Current or past alcohol consumption exceeding 20g/day
* Premature ovarian failure
* History of any active malignancy
* Use of medications known to affect liver enzymes or fat metabolism
* Current participation in another clinical trial

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal women aged 40 years and older were eligible for inclusion. Only biologically female participants were considered, as the study focused on the effects of estrogen deficiency and menopausal hormone therapy.
Enrollment: 44 (Actual)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Change in ATI (Attenuation Imaging) value from baseline to 6 months | Baseline and 6 months
  Quantitative measurement of hepatic steatosis using ultrasound-based attenuation imaging (ATI). A decrease in ATI indicates improvement in hepatic fat content.

SECONDARY OUTCOMES:
Change in FIB-4 Score from baseline to 6 months | Baseline and 6 months
  Assessment of liver fibrosis using FIB-4 score formula: [Age × AST] / [Platelet × √ALT]. Lower scores indicate less fibrosis.
Change in Liver Enzyme Levels (AST, ALT, GGT, LDH) | Baseline and 6 months
  Serum levels of AST, ALT, GGT, and LDH measured through standard laboratory assays to evaluate liver function.
Change in Lipid Profile (LDL, Total Cholesterol) | Baseline and 6 months
  Evaluation of lipid metabolism via total cholesterol and LDL levels to assess metabolic effects of MHT.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University - Cerrahpasa, Cerrahpasa Faculty of Medicine, Istanbul, Beyoğlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
De-identified individual data will be made available upon reasonable request from the corresponding author for academic and non-commercial use.